CLINICAL TRIAL: NCT01297894
Title: Colistin Plus Fosfomycin in Multi-Drug Resistant Acinetobacter Baumannii
Brief Title: Colistin Versus Colistin Plus Fosfomycin for Infections Caused by MDR Acinetobacter Baumannii
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Visanu Thamlikitkul, Division of Infectious Diseases and tropical medicine, Department of medicine, Faculty of Medicine Siriraj Hospital., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Siriraj CEU53-001
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Drug Safety
Keywords: A. baumannii; colistin; fosfomycin
MeSH Terms: interventions — Colistin; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- colistin (Active Comparator): Colistimethate sodium 2.5-5mg/kg iv
  Interventions: Drug: colistin
- colistin plus fosfomycin (Active Comparator): colistimethate sodium 2.5-5mg/kg iv plus fosfomycin 2gm iv every 12 hours
  Interventions: Drug: colistin plus fosfomycin

INTERVENTIONS:
Drug: colistin — Colistimethate sodium 2.5-5mg/kg of colistin base
  Other Names: Colistate
  Arms: colistin
Drug: colistin plus fosfomycin — colitimethate sodium 2.5-5mg/kg iv plus fosfomycin 2gm iv every 12 hours
  Other Names: Colistate; Fosmicin
  Arms: colistin plus fosfomycin

SUMMARY:
In Siriraj Hospital, colistin alone for treatment of MDR A. baumannii contributed to mortality 45% Fosfomycin is an antimicrobial which has activity against gram-negative bacterial including MDR A. baumannii In this study, we compare the clinical and microbiologicalresponse of colistin alone versus colistin plus fosfomycin in treatment of A. baumannii infected patients

DETAILED DESCRIPTION:
Inclusion criteria

* Age> 18 years
* Hospitalized to Siriraj Hospital
* Infected caused by A. baumannii
* Need Colistin treatment

Exclusion criteria

* Pregnancy or Lactating mother
* Colistin or Fosfomycin Allergy
* Patients who have severe abnormal renal or liver function

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Hospitalized to Siriraj Hospital
* Infected caused by A. baumannii
* Need Colistin treatment

Exclusion criteria:

* Pregnancy or Lactating mother
* Colistin or Fosfomycin Allergy
* Patients who have severe abnormal renal or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
number of subjects with cure or improvement | up to 28days
  cure improvement worse death

SECONDARY OUTCOMES:
number of subjects with eradication of causative bacteria | up to 28days
  eradication persistence superinfection

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Sirijatuphat R, Thamlikitkul V. Preliminary study of colistin versus colistin plus fosfomycin for treatment of carbapenem-resistant Acinetobacter baumannii infections. Antimicrob Agents Chemother. 2014 Sep;58(9):5598-601. doi: 10.1128/AAC.02435-13. Epub 2014 Jun 30. PMID 24982065